CLINICAL TRIAL: NCT00444990
Title: A Double-Blind, Randomized, Placebo-Controlled Study on Magnetic Field Therapy to Improve Chronic Lumbar Pain (Lbp)
Brief Title: Study on Magnetic Field Therapy to Improve Chronic Lumbar Pain
Acronym: LBP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Weintraub, Michael I., MD, FACP, FAAN (Individual)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 00781441
Record Dates: First submitted 2007-03-06; First posted 2007-03-08 (Estimated); Last update posted 2007-09-21 (Estimated); Status verified 2007-09

CONDITIONS: Low Back Pain
Keywords: Lumbar pain; magnets; Reduce low back pain
MeSH Terms: conditions — Low Back Pain

INTERVENTIONS:
Device: Magnetic Flex Pad

SUMMARY:
OBJECTIVE:

The objective of this study is to determine if treatment with a flex pad impregnated with static/permanent magnets that can penetrate over 70 mm may improve the quality of chronic lumbar pain with reduction of pain scores.

HYPOTHESIS:

The researchers hypothesis that the application of a flex pad active magnetic therapy vs. sham if utilized daily during waking hours can reduce back pain and/or radicular pain. The null hypothesis is that treatment of subjects with chronic back pain with exposure to static/permanent magnetic fields have no measurable effect on chronic back pain scores and will be equal to the underlying placebo.

DETAILED DESCRIPTION:
DESIGN:

This is a double-blind, randomized, placebo-controlled study which will consist of two treatment groups. Treated subjects will receive a static/permanent magnetic flex pad with a nominal strength of less than 1000 Gauss. Control subjects will receive physically identical flex pad without magnet with a nominal surface field strength of 0 Gauss (placebo). The magnets will be contained in a pad with a Velcro cover and subjects will wear the pad attached to their undergarments/skin during waking hours. Dr. Weintraub will examine participants initially to look for presence or absence of radiculitis, range of motion, presence of absence of spasm, etc. The primary outcome measures will be reduction of chronic low back pain in comparison with prior baseline scores. It is recognized that these changes are subjective in nature. Patients will maintain their VAS scores on a monthly basis and at the end of the study, individuals will return all forms and be reevaluated by Dr. Weintraub. They will be asked specific questions regarding PGIC for bias, etc.

ELIGIBILITY:
Inclusion Criteria:

* Female or male subjects age 18-80.
* Capable of understanding and complying with study protocols.
* Chronic lumbar pain for at least six months

Exclusion Criteria:

* Unable to understand informed consent (mental retardation, psychosis, communicative impairment).
* Cardiac pacemaker or other mechanical internal devices.
* Tumor in the spine/history of malignancy or tumor.
* Pregnancy.
* Prior spine surgery.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-02; Study Completion 2007-12

PRIMARY OUTCOMES:
VAS Pain scores/ SF 15 Pain descriptors/ PGIF/

SECONDARY OUTCOMES:
Autonomic nervous system functions and range of motion

CONTACTS AND LOCATIONS:
Overall Officials: Michael I. Weintraub, MD, Principal Investigator — Phelps Memorial Hospital
Locations (1):
- Michael I. Weintraub, MD, Briarcliff Manor, New York, United States